CLINICAL TRIAL: NCT04883801
Title: Comparison of Early Postnatal Clinical Outcomes of Newborns Born to Pregnant Women With COVID-19: A Case-control Study
Brief Title: Clinical Outcomes of Newborns Born to Pregnant Women With and Without COVID-19
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assistant professor, Kahramanmaras Sutcu Imam University
Other Study IDs: Newborns outcomes
Record Dates: First submitted 2021-05-09; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Vertical Transmission of Infectious Disease; Neonatal Infection; Pregnancy Related
Keywords: Childbirth; COVID-19; Neonatal outcomes; Newborn; Pregnant women; Vertical transmission
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 case group: Newborns born to pregnant women diagnosed with COVID-19 during hospitalization for delivery
  Interventions: Diagnostic Test: Reviewed clinical records and laboratory results
- Control group: Newborns born to pregnant women who were not diagnosed with COVID-19 in their medical history and hospitalization for delivery
  Interventions: Diagnostic Test: Reviewed clinical records and laboratory results

INTERVENTIONS:
Diagnostic Test: Reviewed clinical records and laboratory results — Retrospectively reviewed clinical records and laboratory results

SUMMARY:
A case-control trial was conducted to test the early postpartum period clinical outcomes of newborns born to pregnant women with and without COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women on labor or preterm labor. Pregnant women who underwent programmed or emergence cesarean

Exclusion Criteria:

Those who were transferred to another hospital without or within a short period of delivery

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Newborns born to pregnant women with and without COVID-19 at Denizli State Hospital between March 11, 2020 - March 11, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Vertical transmission | 48 hours after birth
  Determine the prevalence of COVID-19 in newborns born to pregnant women with COVID-19 with PCR from a nasopharyngeal swab.
Neonatal birth outcomes | At birth
  Determine the neonatal outcomes of the newborn specifying the birth week of the newborn, delivery type (vaginal or cesarean), birth weight (g), APGAR scores in the first and fifth minutes after birth.
Neonatal postnatal outcomes | Within 48 hours after birth
  Determine the prevalence of neonatal postnatal outcomes of the newborn specifying the respiratory system illness, intensive care need, oxygen need, neonatal mortality, general health status, and breastfeeding status.

CONTACTS AND LOCATIONS:
Locations (1):
- Denizli State Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No